CLINICAL TRIAL: NCT04509986
Title: GlobalSurg-CovidSurg Week: Determining the Optimal Timing for Surgery Following SARS-CoV-2 Infection
Brief Title: GlobalSurg-CovidSurg Week
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Birmingham (Other)
Collaborators: National Institute for Health Research (NIHR) Global Health Research Unit Grant (NIHR 16.136.79) (Unknown); Association of Coloproctology of Great Britain and Ireland (Unknown); Bowel & Cancer Research (Unknown); Association of Upper Gastrointestinal Surgeons; British Association of Surgical Oncology (Unknown); Bowel Disease Research Foundation (Unknown); British Gynaecological Cancer Society (Unknown); European Society of Coloproctology (Unknown); National Institute for Health Research, United Kingdom (Other Government); Sarcoma UK (Unknown); Vascular Society for Great Britain and Ireland (Unknown); Yorkshire Cancer Research (Other)
Responsible Party: Sponsor
Other Study IDs: GS-CSWeek.20200713
Record Dates: First submitted 2020-08-11; First posted 2020-08-12 (Actual); Last update posted 2020-08-12 (Actual); Status verified 2020-08

CONDITIONS: Surgery; Covid19; Post-Op Complication
MeSH Terms: conditions — COVID-19; Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Observational study to determine the optimal timing for surgery following SARS-CoV-2 infection and assess key global surgery indicators.

DETAILED DESCRIPTION:
* Prospective, observational international cohort study.
* Any hospital worldwide can participate (including hospitals that have not admitted SARS-CoV-2 infected patients).
* All patients undergoing a surgical procedure in an operating theatre will be included. All consecutive eligible patients should be included.
* 7-day data collection period, with follow-up at 30 days after surgery for each patient. However, no changes should be made to normal patient care/ follow-up pathways
* Primary outcome is 30-day mortality.
* All collaborators will be included as PubMed-citable co-authors on resulting publications.

ELIGIBILITY:
Inclusion criteria

* Any operation (elective or emergency) done in an operating theatre by a surgeon.
* All surgical specialties including: acute care surgery, breast surgery, cardiac surgery, colorectal surgery, general surgery, gynaecology, hepatobiliary surgery, neurosurgery, obstetrics, oesophagogastric surgery, ophthalmology, oral and maxillofacial surgery, orthopaedics, otolaryngology, paediatric surgery, plastic surgery, thoracic surgery, transplant surgery, trauma surgery, urology, vascular surgery.
* Day case surgery and inpatient surgery included.
* Any SARS-CoV-2 status (positive at any time, negative, not tested).
* All ages including children and adults.

Exclusion criteria:

Minor procedures (full list will be available in the protocol).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients undergoing surgery done in an operating theatre by a surgeon.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-10-01 (Estimated); Primary Completion 2020-10-31 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
Post-operative mortality | 30 days after surgery
  Mortality at 30 days after surgery

SECONDARY OUTCOMES:
In-patient mortality | 30 days after surgery
  Mortality while the patient is admitted to hospital
Post-operative pulmonary complications | 30 days after surgery
  30-day postoperative pulmonary complications (pneumonia [CDC definition], ARDS, unexpected ventilation)
Post-operative venous thromboembolism | 30 days after surgery
  30-day venous thromboembolism (deep vein thrombosis/ pulmonary embolism)
Post-operative complications | 30 days after surgery
  30-day Clavien-Dindo grade

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] NIHR Global Health Research Unit on Global Surgery; STARSurg Collaborative. A prognostic model for use before elective surgery to estimate the risk of postoperative pulmonary complications (GSU-Pulmonary Score): a development and validation study in three international cohorts. Lancet Digit Health. 2024 Jul;6(7):e507-e519. doi: 10.1016/S2589-7500(24)00065-7. PMID 38906616
- [Derived] Glasbey J; COVIDSurg and GlobalSurg Collaboratives. Peri-operative outcomes of surgery in children with SARS-CoV-2 infection. Anaesthesia. 2022 Jan;77(1):108-109. doi: 10.1111/anae.15614. Epub 2021 Nov 5. No abstract available. PMID 34739137
- [Derived] Nepogodiev D; COVIDSurg and GlobalSurg Collaboratives. Timing of surgery following SARS-CoV-2 infection: country income analysis. Anaesthesia. 2022 Jan;77(1):111-112. doi: 10.1111/anae.15615. Epub 2021 Nov 5. No abstract available. PMID 34739085
- [Derived] Lobo D, Devys JM. Timing of surgery following SARS-CoV-2 infection: an international prospective cohort study. Anaesthesia. 2022 Jan;77(1):110. doi: 10.1111/anae.15540. Epub 2021 Jul 12. No abstract available. PMID 34251685
- [Derived] COVIDSurg Collaborative, GlobalSurg Collaborative. SARS-CoV-2 vaccination modelling for safe surgery to save lives: data from an international prospective cohort study. Br J Surg. 2021 Sep 27;108(9):1056-1063. doi: 10.1093/bjs/znab101. PMID 33761533